CLINICAL TRIAL: NCT00744120
Title: Lymphoma Follow-up Protocol
Brief Title: Lymphoma Follow-up
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: AG0108
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Lymphoma
Keywords: cancer
MeSH Terms: conditions — Lymphoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This follow-up protocol is designed to evaluate participants who have previously been lymphoma patients treated on approved clinical studies of the National Institutes of Health.

DETAILED DESCRIPTION:
The intent of this protocol is to accrue up to 800 volunteers who are interested in participating in NIA research studies as part of follow-up for previous cancer treatment at NIH. Participants will be asked to answer questions regarding their general health status, diagnoses, and admissions to hospital, and to provide possible documentation. They may be asked to come to the NIA Clinical Research Unit at Harbor Hospital to participate in a follow-up evaluation. They will have the opportunity to obtain additional information about studies in which they may wish to participate and to discuss eligibility issues with NIA staff members. Any identified clinical problems in need of care will also be discussed. Volunteers may be referred, with their permission, to their private medical doctor for follow-up. They may be re-evaluated within a year for further follow-up.

The follow-up evaluation may include history and physical, blood and urine tests, questionnaire, MRI or CT.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated on an approved NCI/NIH protocols
* Willing and able to provide informed consent for current NIA protocol
* Rare, unusual, interesting or unknown condition that requires diagnosis

Exclusion Criteria:

* Does not meet the criteria of any previously-approved NIH Protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, previously entered on NIH study who may be eligible if they have rare, unusual, interesting or unknown conditions that require diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2003-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Long-term survival following treatment for lymphoma | Annually

SECONDARY OUTCOMES:
Long-term toxicity possibly attributable to lymphoma or treatment for lymphoma | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L. Duffey, RN, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- NIA Clinical Research Unit, Baltimore, Maryland, United States